CLINICAL TRIAL: NCT03926351
Title: A Randomized, 24 Week Parallel-group Placebo-controlled (Phase 2) Pilot-study of High Dose Omega 3 (DHA) in People at Risk for Dementia
Brief Title: High Dose Omega 3 in People at Risk for Dementia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: BASF AS (Industry); Pre Diagnostics (Industry)
Responsible Party: Principal Investigator, Nora Christine Lund Sørbøe, research fellow, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REC: 2017/1364
Record Dates: First submitted 2019-03-11; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Dementia; Inflammation; Mild Cognitive Impairment; Cognitive Decline; SCD; Cognitive Dysfunction; Pathologic Processes; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorder; Cognition Disorders
MeSH Terms: conditions — Dementia; Inflammation; Cognitive Dysfunction; Pathologic Processes; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorders; Cognition Disorders | interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Intervention Model Description: A randomized, 24-week parallel-group placebo-controlled (Phase 2) pilot-study of high dose Omega 3 (DHA) in people at risk for dementia
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1a; Placebo (Placebo Comparator): Valid for the first 24 weeks of the study. Arm 1a: placebo, soft gelatine capsule containing 1000 mg olive oil, refined.
  Interventions: Dietary Supplement: Olive oil
- Arm 2a; Omega-3 capsules (Experimental): Valid for the first 24 weeks of the study. Arm 2a; Omega-3, (1000 mg fill weight per capsule) containing omega-3 ethyl ester concentrate with a high proportion of DHA.
  Interventions: Dietary Supplement: Omega-3 capsules

INTERVENTIONS:
Dietary Supplement: Omega-3 capsules — BASF AS is the developer of the gelatine capsules containing Omega-3 ethyl ester from fish oil concentrate, as the dietary (nutritional) ingredient. The additional capsule fill ingredients are food additives permitted in food supplements according to Regulation (EC) No 1333/2008 on Food additives.
  Arms: Arm 2a; Omega-3 capsules
Dietary Supplement: Olive oil — Soft gelatine capsule containing 1000 mg olive oil, refined.
  Arms: Arm 1a; Placebo

SUMMARY:
The aim of this study is the efficacy of a docosahexaenoic acid (DHA)-rich dietary supplement in improving key dementia-related mechanisms and cognitive function in older people at risk for dementia. This is a randomized placebo-controlled, 24 weeks, phase 2 study of Omega 3 in people with increased risk of dementia. The aim is to explore the effects of DHA on cognitive performance (CERAD 10 word memory tests, TMT A/B, Stroop Color-Word, FAS, VOSP silhouettes, Cantab-test (RT, PAL, SWT)), biological markers (blood: CRP, NLF, TNF-alpha, MCI-1, PBMC Abeta middomain, Omega-3-index, IL, CSF: NLF, sTREM2, Ab 1-42, total and -phospho-tau) and imaging (MRI: standard structural DDI protocol including Freesurfer and WML measurements, DTI and ASL).

DETAILED DESCRIPTION:
Earlier trials with eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) have been moderately promising, but these interventions often suffered from relatively low DHA concentrations. In this trial, the investigators will use a DHA-rich dietary supplement formulated using a self-microemulsifying delivery system to accelerate absorption.

Modification of innate immune activity has already been seen using DHA-rich supplements, and this type of intervention has been shown to ameliorate AD-associated PBMC profiles, and to be associated with improvements in cognition. DHA can cross the BBB, and the resulting CSF concentrations are associated with reduced CSF total tau levels indicating that DHA reduce neurodegeneration, ameliorate Abeta42 induced neuronal damage, and increase microglia Abeta phagocytosis. However, pre-clinical and pre-dementia intervention trials linked to biomarkers for the AD disease process is lacking, and therefore, stratification with respect to stage of disease process has not been performed.

Study cohort: subjects in this pilot study will be recruited from the Norwegian Dementia Disease Initiative (DDI) cohort. The DDI cohort consists of 600 participants with Subjective Cognitive Dedcline (SCD), Mild Cognitive Impairment (MCI) and normal control subjects that have been included at dementia centres across Norway during 2012-2016. Blood samples and cerebrospinal fluid (CSF) have been collected and are stored centrally at Ahus. A comprehensive and highly standarized clinical assessment program has been administered by trained raters (assessors). The investigators are currently performing 2-year follow-up evaluations. Genetic data including APOE-isoforms have been collected as have baseline and follow-up MRIs, PET scans (so far in Oslo and Bergen) and baseline CSF examinations (Ab, total-tau and phosphorus-tau). Cognitive assessments at baseline and follow-up include MMSE and Clinical Dementia Rating (CDR), CERAD 10 word memory test, Clock drawing test, Trail Making Test A and B, Verbal fluency test (FAS), visual recognition test (VOSP silhouettes), Stropp Coloraturas-Word. Data is assembled in a customised database (UiO secure server (TSD)), developed based on XNAT (http://www.xnat.org) and also connected to pipelines for image analysis. A selection from CANTAB MCI test battery including RTI (reaction time), PAL (paired associates learning test), and SWM (spatial working memory).

Study design: All subjects included in the intervention study will have completed 2-year follow-up in the DDI study prior to inclusion and will be on stable medication at least 3 months prior to baseline examinations. Based on the existing electronic CRF for DDI, social e-RCT-CRFs will be developed and programmed into the proprietary XNAT database. Patients fulfilling the inclusion criteria will be identified by a nurse at the memory outpatient clinics and will be given a short information letter regarding the study. Written consent will be asked for. Thereafter, a medical and neurological examination of the patient will be performed, including a medical history and medication use.

This initial pilot study is a minor feasibility study with 40 subjects randomised equally to either of 2 treatment groups for 24 weeks,

Omega-3 3 capsules/day Placebo 3 capsules/day

Each study participant will take 3 capsules in the morning for the 24-week study period. The study may be followed by a larger and statistical valid study. Patients will be randomized (by means of a computerized program) to identically appearing set of capsules with Omega-3 or placebo, 1:1 (produced by BASF AS).

Optional extension study: Participants will be offered another 24-week Omega-3 capsule supply after study end, and a follow-up assessment after 1 year will be conducted, comparing those with and without continuous Omega-3 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* SCD or MCI
* No evidence of neurodegeneration (i.e. CSF phospho and total tau-levels below cut-off)
* Scandinavian mother tongue
* Completed 2-year follow-up in the DDI-study
* Stable medication for at least 3 months prior to baseline exam

Exclusion Criteria:

* Dementia (defined as MMSE < 26 and/or CDR >/= 1))
* Other dementia giving disease than AD
* Other brain disease
* Significant depression
* Unstable coronary heart disease or heart failure in need of treatment
* Systemic inflammatory diseases
* Somatic disease that might affect cognitive function adversely
* Usage of anticoagulants
* Prior radiation- or chemo-therapy possibly affecting CNS
* Relevant cancer or other serious disease with expected survival < 5 years
* Fish meal intake more than 2 times a week
* Regularly intake of Omega-3 supplements over the last 3 months

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | Baseline to 24 weeks
  CERAD 10 word memory test relative to placebo

SECONDARY OUTCOMES:
Cognitive function | Baseline to 24 weeks
  Cantab RT test relative to placebo
Cognitive function | Baseline to 24 weeks
  Cantab PAL test relative to placebo
Cognitive function | Baseline to 24 weeks
  Cantab SWT test relative to placebo
Blood PBMC betaAmyloid mid-domain assay | Baseline to 24 weeks
  IVD assay
CSF betaAmyloid 1-42 | Baseline to 24 weeks
  IVD assay
CSF TAU | Baseline to 24 weeks
  IVD assay
CSF Phospho-TAU | Baseline to 24 weeks
  IVD assay
MRI ASL | Baseline to 24 weeks
  MRI procedure
MRI WML | Baseline to 24 weeks
  MRI procedure
MRI DTI | Baseline to 24 weeks
  MRI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Tormod Fladby, MD PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus university hospital, Sykehusveien 25, Lørenskog, Norway